CLINICAL TRIAL: NCT03618628
Title: Carbon Fiber Off-Loading Orthosis
Brief Title: Peak Plantar Pressures While Wearing a Carbon Fiber Off Loading Orthoses
Acronym: CFO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Mary Hastings, PT, DPT, ATC, Professor of Physical Therapy, Orthopaedic Surgery, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201308105
Record Dates: First submitted 2018-07-16; First posted 2018-08-07 (Actual); Results first posted 2019-05-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Diabetes Mellitus; Peripheral Neuropathy; Orthotic Device
MeSH Terms: conditions — Diabetes Mellitus; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- People using a CFO (Experimental): People who are currently wearing a carbon fiber off loading orthosis (CFO) will have a new CFO fabricated for them based on the results of our finite element (FE) model. We will then test both CFOs ability to reduce peak plantar compared to barefoot and the peak plantarflexor power of both braces.
  Interventions: Device: Carbon Fiber Off Loading Orthosis (CFO)

INTERVENTIONS:
Device: Carbon Fiber Off Loading Orthosis (CFO) — A finite element (FE) model will be created to determine properties that will improve CFO strength while maintaining reduction of peak plantar pressures of the CFO and plantarflexor power. A new CFO will then be fabricated for the participant. Participants will be tested in while walking barefoot, wearing their current CFO, and wearing the FE model driven CFO.

SUMMARY:
The purpose of this study is to determine the ability of carbon fiber off loading orthoses to reduce plantar pressure while providing an augmented plantarflexor power to improve walking and function. Results of this study could lead to increased use of carbon fiber off loading orthoses for patients with diabetes, peripheral neuropathy, and foot wounds as a way augmenting wound healing and preventing future recurrences of wounds.

DETAILED DESCRIPTION:
The long term goal of this research is the successful incorporation of carbon fiber into an off loading device will provide protection to the insensate foot of people with diabetes by reducing localized peak pressures, and thus the risk of recurrence neuropathic foot wounds and fractures, while improving ankle power at push off that will allow individuals with loss of ankle muscle function to walk faster and return to dynamic activities required in their jobs and for full function in the community. The overall goal of this proposal is to determine effects of carbon fiber off loading orthoses (CFO) design characteristics (lay up and geometry of strut) on brace strength, weight, power return capacity, plantar off-loading and participant comfort using FE models, ex-vivo testing and human testing.

First, a CFO will be fabricated using geometry consistent with the current clinical standard. This representative CFO will serve as a baseline from which a finite element (FE) model will be built. The model will be altered as desired to determine the effects of variable design characteristics. The FE model will estimate brace deflection and stress when the CFO is designed with various lay up designs and brace thicknesses. We will use results from the FE model to fabricate a new CFO for study participants.

We will then measure peak plantar pressures during walking while the participants are barefoot, wearing the CFO consistent with current clinical standards, and wearing the new CFO fabricated based on the results of the FE model. We will also measure plantarflexor power during walking while the participants are wearing the CFO consistent with current clinical standards and while wearing the CFO designed based on the results of the FE model. It is believed that the FE model driven CFO design will lead to improved brace strength while reducing plantar pressure compared to barefoot and will have similar plantarflexor power as the CFO based on current clinical standards.

ELIGIBILITY:
Inclusion Criteria:

1. Daily life includes a minimum of moderate activity level (variable cadence walking)
2. Have a Gillette or carbon off loading orthosis as a result of diabetes related foot impairments
3. Diagnosis of diabetes mellitus and peripheral neuropathy
4. Ability to ambulate in the community (K-level ≥ 2)
5. Age > 21 years

Exclusion Criteria:

1. Unable to ambulate and complete testing required for study participation.
2. Severe foot deformity of the hindfoot or any deformity of the foot with a dislocation resulting in a bony prominence on the plantar/weightbearing surface of the foot.
3. Neurological diseases that affects walking

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2018-04-12 (Actual); Study Completion 2018-04-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary Hastings, DPT, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | People Using a CFO
Started | 3
Completed | 1
Not Completed | 2
Not completed — Death | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | People Using a CFO
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Peak Plantar Pressure
Description: Plantar pressure during walking while the participant wears the brace fabricated based on the finite element (FE) model compared to 1) the brace fabricated based on current clinical standards and 2) barefoot.
Time Frame: Participant was tested in new brace (based on FE model) after wearing for 1 week.
Measure: Number; unit: Newtons per squared centimeters
Arm/Group | People Using a CFO
Number analyzed (Participants) | 1
Newtons per squared centimeters
  Barefoot (midfoot) | 75.3
  Current CFO (midfoot) | 14.2
  Model driven CFO (midfoot) | 14.5
  Barefoot (Forefoot) | 22.8
  Current CFO (Forefoot) | 3.5
  Model driven CFO (Forefoot) | 6.6
  Barefoot (Heel) | 60.0
  Current CFO (Heel) | 23.4
  Model driven CFO (Heel) | 14.5

ADVERSE EVENTS:
Time Frame: Baseline data collected in a brace provided as standard of care. A finite element model was constructed of the brace and provided input for changes in brace construction. This process took 9 months and the participant was tested in the model informed brace 11 months after initial testing
Description: Risks to participants were the possibility of discomfort, blister, or sore while getting used to a new brace and falling during peak plantar pressure testing. Participants were told to contact the study team immediately if any of these they experienced discomfort, blisters, or sores when adapting to the new brace. During peak plantar pressure testing a study team member walked beside the participant holding a gait belt around the waist to make sure they did not fall.
Arm/Group | People Using a CFO
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT03618628/Prot_SAP_ICF_000.pdf